CLINICAL TRIAL: NCT06705998
Title: A Phase I, Two Parts Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of BAR502 in Healthy Subjects
Brief Title: To Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BAR502 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BAR Pharmaceuticals s.r.l. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: BAR-502-001
Record Dates: First submitted 2024-08-23; First posted 2024-11-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: NASH
Keywords: Non-alcoholic Fatty Liver DIsease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — BAR502

STUDY DESIGN:
Intervention Model Description: The Part A of the study follows a randomised, double-blind, placebo-controlled, parallel group design. The participants are enrolled in 4 consecutive cohorts of 8 healthy subjects each. In each cohort, the first 2 groups include 2 subjects each, while the 3rd group in each cohort includes 4 subjects. Each group of subjects is exposed to the treatment under investigation only if the Investigator's evaluation of the previous group's safety data up to 72 h post-dose is satisfactory and if the competent Ethics Committee gives written authorisation to continue with the next group. At the end of each cohort, before proceeding to the next dose level, safety and tolerability results up to 168 h post-dose (Day 8) are evaluated by a Data Safety Monitoring Board.
  Part B of the study: Two ascending doses of IMP identified in study Part A, are subsequentially administered as daily multiple doses for 2 consecutive weeks (14 days) in two cohorts of 10 healthy subjects each.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind: Active or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAR502 single dose (Experimental): Each subject will receive an oral single-dose of BAR 502 [Study Part A]
  Interventions: Drug: BAR502 single dose
- Placebo single dose (Placebo Comparator): Each subject will receive an oral single-dose of placebo [Study Part A]
  Interventions: Drug: Placebo single dose
- BAR502 multiple doses (Experimental): Each subject will receive a dose of BAR502 once a day for 14 days [Study Part B]
  Interventions: Drug: BAR502 multiple doses

INTERVENTIONS:
Drug: BAR502 single dose — Single oral doses of BAR 502/placebo will be administered as film-coated tablets, in the morning of Day 1, with 150 mL of water, after an overnight fasting of at least 8 hours.
  BAR 502 film-coated tablets are available at dose strengths of 3, 10 and 50mg. A maximum of 4 dose levels are pre-planned (3, 10, 30 and 60mg).
  Arms: BAR502 single dose
Drug: Placebo single dose — Matching BAR 502 placebo film-coated tablets will be given to 2 out of 8 subjects in each cohort using the same regimen as outlined for the active study treatment
  Arms: Placebo single dose
Drug: BAR502 multiple doses — The 2 multiple ascending doses selected based on results of study part A will be administered to 2 study cohorts of 10 subjects each. The IMP will be orally administered once a day from Day 1 to Day 14, at 8:00±1 h, for a total of 14 doses.
  Arms: BAR502 multiple doses

SUMMARY:
First-in-human, single centre, two parts, dose-escalation, parallel-group, safety, tolerability, pharmacokinetic and pharmacodynamic Phase I study. Part A: randomised, double-blind, placebo-controlled, single ascending dose study.

Part B: open label, multiple ascending dose study.

DETAILED DESCRIPTION:
First-in-human, single centre, two parts, dose-escalation, parallel-group, safety, tolerability, pharmacokinetic and pharmacodynamic Phase I study. Part A: randomised, double-blind, placebo-controlled, single ascending dose study to evaluate the safety and tolerability of BAR502 and matching placebo across 4 single ascending doses administered to 4 cohorts of 8 healthy subjects each.

Part B: open label, multiple ascending dose study to evaluate the safety and tolerability of two ascending doses of BAR502, considered as safe in study Part A, when administered as multiple doses to 2 cohorts of 10 healthy subjects each.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: men/women, 18-55 years old inclusive
3. Body Mass Index: 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-99 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
6. Renal functionality: estimated glomerular filtration rate calculated using the Cockcroft-Gault equation and normalized to an average surface area of 1.73 m2 ≥ 90 mL/min at screening
7. Tobacco: non-smokers, non-users of nicotine containing products and non-users of Vapo e-cigarettes for at least 3 months prior to study screening
8. Contraception and fertility (women only): women of non-child-bearing potential or in post-menopausal status for at least 1 year, defined as such when there is either:

   1. 12 months of spontaneous amenorrhea or
   2. 6 weeks documented postsurgical bilateral oophorectomy with or without hysterectomy will be admitted. For all women, pregnancy test result must be negative at screening and on Day -1 of each study part.
9. Contraception (men only): men will either be sterile or agree to use one of the following approved methods of contraception from the first investigational medicinal product administration until at least 90 days after the last administration, also in case their partner is currently pregnant:

   1. A male condom with spermicide
   2. A sterile sexual partner or a partner in post-menopausal status for at least 1 year
   3. Use by the female sexual partner of an IUD, a female condom with spermicide, a contraceptive sponge with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, or hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit or: True abstinence

Exclusion Criteria:

1. ECG 12-leads (supine position): clinically significant abnormalities, in particular QTcF > 450 ms
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values at screening indicative of physical illness or any acute laboratory abnormality at Screening which, in the opinion of the Investigator, should preclude participation in the study of an investigational compound. INR > 1.2
4. Diseases: significant history of renal, hepatic (in particular, liver or hepatobiliary diseases as indicated by serum alanine aminotransferase, aspartate aminotransferase or total bilirubin levels exceeding the upper limit of normality), gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
5. Gallbladder: history of cholecystectomy, presence of gallstones or clinically significant gallbladder abnormalities that may interfere with the aim of the study
6. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
7. Medications: medications, including over the counter medications, homeopathic preparations, vitamins, food supplements and herbal remedies for 3 weeks before the start of the study
8. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
9. Blood donation: blood donations for 3 months before this study
10. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for men, defined according to the USDA Dietary Guidelines 2020-2025] or caffeine (>5 cups coffee/tea/day) abuse
11. SARS-CoV-2 test: positive Covid-19 rapid test at Day -1
12. Cotinine: positive cotinine test at screening
13. Drug test: positive result at the urine drug screening test at screening or Day -1
14. Alcohol test: positive alcohol saliva test at screening or Day -1
15. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians and vegans
16. Pregnancy (women only): positive or missing pregnancy test at screening or Day -1; child-bearing potential, pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | PART A: Day-15/-2; Day-1 to Day4; Day 8; Day15 - PART B: Day-15/-2 to Day18; Day30
  Safety will be evaluated through the assessment of adverse events
Change in vital sign - BP | PART A: Day-1 to Day4; Day 8; - PART B: Day-15/-2 to Day15; Day18
  Tolerability will be evaluated throught the change in Blood preassure from baseline
Change in vital sign - HR | PART A: Day-1 to Day4; Day 8; - PART B: Day-15/-2 to Day15; Day18
  Tolerability will be evaluated throught the change in Heart rate from baseline

SECONDARY OUTCOMES:
Plasma BAR502 - Study Part A | Day1 (pre- and post- dose), Day2, Day3, Day4
  Plasma BAR502 concentration-time profile after IMP single dose administration
Urine BAR502 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 concentration-time profile after IMP single dose administration
Plasma BAR505 - Study Part A | Day1 (pre- and post- dose), Day2, Day3, Day4
  Plasma BAR505 concentration-time profiles after IMP single dose administration
Urine BAR505 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR505 concentration-time profiles after IMP single dose administration
Plasma BAR502 PK: Cmax - Study Part A | Day1 (pre- and post- dose), Day2, Day3, Day4
  Plasma BAR502 Cmax value after IMP single dose administration
Plasma BAR502 PK: t_max - Study Part A | Day1 (pre- and post- dose), Day2, Day3, Day4
  Plasma BAR502 t_max value after IMP single dose administration
Plasma BAR502 PK: AUC0-t - Study Part A | Day1 (pre- and post- dose), Day2, Day3, Day4
  Plasma BAR502 AUC0-t value after IMP single dose administration
Urine BAR502 PK: Ae0-t - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 Ae0-t value after IMP single dose administration
Urine BAR502 PK: Fe0-t - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 Fe0-t value after IMP single dose administration
Urine BAR502 PK: Rmax - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 Rmax value after IMP single dose administration
Urine BAR502 PK: AUR_Clast - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 AUR_Clast value after IMP single dose administration
Urine BAR502 PK: REC% - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 REC% value after IMP single dose administration
Urine BAR502 PK: tu_max - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 tu_max value after IMP single dose administration
Urine BAR502 PK: Cl_r r - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Urine BAR502 Cl_r r value after IMP single dose administration
Serum biomarker FGF19 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum FGF19 baseline-corrected concentration-time profile after IMP single dose administration
Serum biomarker C4 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum C4 baseline-corrected concentration-time profile and PD parameters after IMP single dose administration
Serum biomarker GLP-1 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum GLP-1 baseline-corrected concentration-time profile after IMP single dose administration
Serum PD: Cb_max - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum Cb_max value after IMP single dose administration
Serum PD: Cb_min - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum Cb_min value after IMP single dose administration
Serum PD: tb_max - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum PD tb_max value after IMP single dose administration
Serum PD: tb_min - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum tb_min value after IMP single dose administration
Serum PD: AUbC_0-24 - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum AUbC_0-24 value after IMP single dose administration
Serum PD: partial AUbC - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum partial AUbC value after IMP single dose administration
Serum total bile acids - Study Part A | Day1 (pre- and post- dose), Day2, Day3
  Serum total bile acids baseline-corrected concentration-time profiles after IMP single dose administration
Plasma BAR502 concentration - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR502 concentration-time profile after IMP multiple dose
Plasma BAR505 concentration - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR505 concentration-time profile after IMP multiple dose
Plasma BAR502 PK: Cmax - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR502 Cmax value after IMP multiple dose
Plasma BAR502 PK: t_max - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR502 t_max value after IMP multiple dose
Plasma BAR502 PK: AUC_0-24 - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR502 AUC_0-24 value after IMP multiple dose
Plasma BAR502 PK: AUC_0-t - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day18
  Plasma BAR502 AUC_0-t value after IMP multiple dose
Serum biomarker GLP-1 - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum GLP-1 baseline-corrected concentration-time profile after IMP multiple dose
Serum biomarker C4 - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum C4 baseline-corrected concentration-time profile after IMP multiple dose
Serum biomarker FGF19 - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum FGF19 baseline-corrected concentration-time profile after IMP multiple dose
Serum PD: Cb_max - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum Cb_max value after IMP multiple dose
Serum PD: Cb_min - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum Cb_min value after IMP multiple dose
Serum PD: tb_max - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum tb_max value after IMP multiple dose
Serum PD: tb_min - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum tb_min after IMP multiple dose
Serum PD: AUbC_0-24 - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum AUbC_0-24 value after IMP multiple dose
Serum PD: partial AUbC - Study Part B | daily from Day1 to Day14 (pre- and post- dose); Day15 to Day17
  Serum partial AUbC value after IMP multiple dose
Serum total bile acids - Study Part B | Daily from Day1 to Day17
  Serum total bile acids baseline-corrected concentration-time profiles after after IMP multiple dose
Change in body weight | PART A: Day1; Day 8 - PART B: Day1; Day18; Day30
  Change in body weight from baseline after single and multiple IMP dose
Check for Physical abnormalities | PART A: Day1; Day 8 - PART B: Day1; Day18; Day30
  Change in Physical examination from baseline after single and multiple IMP dose
hepatic parameters: AST | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in AST value after single and multiple IMP dose
hepatic parameters: ALT | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in ALT value after single and multiple IMP dose
hepatic parameters: Total bilirubin | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in Total bilirubin value after single and multiple IMP dose
hepatic parameters: Direct bilirubin | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in Direct bilirubin value after single and multiple IMP dose
hepatic parameters: Indirect bilirubin | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in Indirect bilirubin value after single and multiple IMP dose
hepatic parameters: Total cholesterol | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in Total cholesterol value after single and multiple IMP dose
hepatic parameters: HDL cholesterol | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in HDL cholesterol value after single and multiple IMP dose
hepatic parameters: LDL cholesterol | PART A: Day2; Day3; Day 8; - PART B: daily from Day2 to Day13; Day15; Day18
  Change from baseline in LDL cholesterol value after single and multiple IMP dose
Change in Gallbladder contraction - Study Part B | daily from Day2 to Day13; Day15
  Change from baseline in Gallbladder contraction after IMP multiple dose
Change in Gallbladder volume - Study Part B | daily from Day2 to Day13; Day15
  Change from baseline in Gallbladder volume after IMP multiple dose
Change in ECG trace: PR | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG trace PR interval value after single and multiple IMP dose
Change in ECG trace: QRS | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG trace QRS interval value after single and multiple IMP dose
Change in ECG trace: QT | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG trace QT interval value after single and multiple IMP dose
Change in ECG trace: QTcB | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG trace QT interval corrected with Bazett's formula after single and multiple IMP dose
Change in ECG trace: QTcF | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG trace QT interval corrected with Fridericia's formula after single and multiple IMP dose
Change in ECG: Heart rate | PART A: daily from Day1 to Day 4 - PART B: daily from Day to Day15
  Change from baseline in ECG Heart rate after single and multiple IMP dose

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A., Phase I Unit
Locations (1):
- CROSS Research S.A. Phase I Unit, Arzo, Switzerland

IPD SHARING:
Plan to Share IPD: No